CLINICAL TRIAL: NCT01557023
Title: Clinical Trial With Combination of Dienogest/Ethytnilestradiol and Drosperidona/Ethyniestradiol
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Change Company strategy
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EF 124 NINA
Record Dates: First submitted 2012-03-08; First posted 2012-03-19 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2012-03

CONDITIONS: Metrorrhagia
MeSH Terms: conditions — Metrorrhagia | interventions — Contraception, Barrier

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dienogest 2 mg/ethynilestradiol 30 mcg; (Experimental)
  Interventions: Drug: barrier methods
- Yasmin® (Active Comparator)
  Interventions: Drug: barrier methods

INTERVENTIONS:
Drug: barrier methods
  Arms: dienogest 2 mg/ethynilestradiol 30 mcg;
Drug: barrier methods
  Arms: Yasmin®

SUMMARY:
This trial will study the percentage of women with at least one occurrence of intracyclic bleeding (bleeding and/or spotting) during the cycles 2 and 3 of treatment with test or reference drug.

ELIGIBILITY:
Inclusion Criteria:

* Sign, initial and date the informed consent form;
* Female patients, with child bearing potential, aged 18 to 35 years;
* Have indication to receive progesterone and estrogen-based low oral hormone treatment for at least 7 cycles (approximately 7 months) for birth control;
* Be able to comply with the study protocol;
* Show normal result in cervical-vaginal cytology conducted up to 3 months before study enrollment or be willing to repeat the screening visit test, which result must also be normal;
* Be willing to use one of the study drugs

Exclusion Criteria:

* Is pregnant or breastfeeding, suspecting to be or planning to get pregnant;
* Patients currently using oral contraceptives with drospirenone 3 mg/ ethynilestradiol 30 mcg or dianogest 2 mg/ ethynilestradiol 30 mcg.
* Have history of gynecologic surgery such as hysterectomy, total oophorectomy or tubal ligation;
* Smoke over 10 cigarettes a day;
* Have any severe comorbidities (at the investigator's criteria), including bowel inflammatory disease
* Have hypertension, showing at least one of the following conditions:

Systolic pressure >140 mm Hg or diastolic pressure >90 mm Hg in sitting position;

* Current use of pharmacological treatment for hypertension;
* Show history or currently have venous or arterial thromboembolism;
* History of breast or genital cancer;
* Have obesity (BMI >30 kg/m2);
* Have liver disease or changed lab values;
* Currently have dysplasia or malignancy in cervical-vaginal cytology;
* Concomitantly use CYP3A4 metabolizing drugs or drugs causing drug interaction with other study drugs;
* History of abortion one (1) month before study enrollment;
* History of childbirth or breastfeeding 3 months before study enrollment;
* Have hypersensitivity to any of the study drug components;
* Patients with long-term disability, who have undergone a major surgery or any surgery in legs or major traumatism in the last 6 months;
* Have current diagnosis of sexually transmitted disease;
* Have used injectable hormones 3 months before study enrollment;
* Have used hormone implant 6 months before study enrollment;
* Have participated in another clinical trial in the last 12 months.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07-01 (Estimated); Primary Completion 2014-12-01 (Estimated); Study Completion 2014-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of intracyclic bleeding and/or spotting during the cycles 2 and 3 of treatment | 2 and 3 cycles (each cycle is 21 days)

SECONDARY OUTCOMES:
Percentage of women with intracyclic bleeding during treatment cycles 2 to 7 | 2 and 7 cycles (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Saúde e Bem Estar da Mulher, São Paulo, Brazil